CLINICAL TRIAL: NCT06916260
Title: Light Therapy Intervention in Individuals With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: NeuroThera (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2277769
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: There will be two groups that receive the light therapy and two that ill receive a placebo treatment to control for any possible effects of the therapy.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Light therapy grpup (Active Comparator)
  Interventions: Device: Red Light (PDT)
- placebo light therapy (Sham Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Red Light (PDT) — The intervention is a non invasive and safe practice. By delivering low level wavelength red light to the front part of the head, it can increase blood flow in the area treated and improve functioning of the associated regions, potentially improving symptoms.
  Arms: Light therapy grpup
Device: Placebo — The intervention is a non invasive and safe practice. Participants will be wearing a helmet that delivered low level light therapy to the brain, and use it for the same amount of time as the treatment group. These participants will however, not receive the actual light and receive a placebo, so the helmet will be off. This is done to control of any potential positive effects of the therapy.
  Arms: placebo light therapy

SUMMARY:
The study looks to investigate the effects that light therapy delivered to the frontal cortex could have on Parkinson's disease related symptoms ( both cognitive and motor). The therapy is a non invasive technique that deliverers low level wavelength light to the front part of the head for 12 minutes. for this study the therapy will be done 3 times a week for 6 weeks. To measure the potential effects on the therapy in Parkinson symptoms, we will do a set of cognitive and motor test before and after the intervention to measure any changes as well as control for any potential markers such as age, sex, disease level, medication and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson disease

Exclusion Criteria:

1. Participants who are unable to comply with study visit/testing requirements (e.g.

   participants who cannot go off PD medication for the pre-, post-, and 3-month assessments).
2. Participants who are unable to provide consent.
3. Participants with a Deep Brain Stimulation (DBS) device.
4. Participants who have a history of a psychiatric disorder
5. Participants with PD who have other concurrent movement/neurological conditions, including dystonia, dementia, epilepsy etc.
6. Participants with a clinical diagnosis of PD that is not considered primary (e.g.

   vascular parkinsonism) or participants where an atypical form of parkinsonism is suspected (e.g., progressive supranuclear palsy, multiple system atrophy).
7. Participants with a history of cancer (whether treated with chemotherapy and/or radiotherapy or not).
8. Participants with a history of a recent concussion or any facial, neck, or head injury within the last 6 months. UD IRB Approved: 03/12/2025 IRBNet ID#: 2277769-2 I/C from Rev. 01/2024 Page 3 of 10 Participant's Initial's ________
9. Known injury or disease that might interfere with motor function in the proposed experiments (e.g., stroke, traumatic brain injury, extrapyramidal dysfunction, neuromuscular disease, orthopedic problems that impair movement).
10. Participants with a history of photosensitivity.
11. Participants who are not able to walk unassisted for 2 minutes

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-04 (Estimated); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
cognitive symptom improvement | Done immediately before (pre test) and after (post test) intervention lasting about 1 hour. The intervention lasts about 6 weeks, so in between the pre and post tests there will be about a 6 week period.
  The investigators want to asses whether light therapy has a positive effect on reducing the cognitive symptoms related with PD, such as loss of short term memory, attention and processing speed. This will be measured using a set of tests and questioners (i.e MoCa, NIH cognitive battery, brief Test of attention (BTA)). Performance on these tests and questioners, which measure diverse aspects of cognition, will be compared before and after the intervention to establish if there is a positive effect of the therapy on any aspect of cognition. The intervention will last a total of 6 weeks right after the completion of the pre intervention assessment. after the completion of the 6 weeks of intervention therapy, the pre test will be conducted and cognitive measure changes will be recorded.
motor symptoms | Done immediately before (pre test) and after(post test) intervention lasting about 1 hour. The intervention lasts 6 weeks, so there is about a 6 week period in between the two sessions ( pre and post)
  The investigators want to asses whether light therapy has a positive effect on reducing the motor symptoms related with PD, such as changes in gait, tremors, and slowing of movement. This will be measured using a set of tests and questioners (i.e MDSUPDRS, Dual task walking, APDM motion capture over a set of tests). Performance on these tests and questioners, which measure diverse aspects of motor capabilities, will be compared before (pre test) and after (post tests) the intervention to establish if there is a positive effect of the therapy on any aspect of motor control and movement. The intervention will last a total of 6 weeks, done right after the completion of the pre intervention assessment. after the completion of the 6 weeks of intervention therapy, the pre test will be conducted and any changes in motor measures will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware STAR Tower, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No